CLINICAL TRIAL: NCT03069417
Title: Project INSPireD: Integrating Nuanced Support for Perinatal Adherence and Depression
Brief Title: Support for Perinatal Adherence and Depression
Acronym: INSPireD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Match Research (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Christina Psaros, Assistant Professor of Psychology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016P001887; K23MH096651 (NIH)
Record Dates: First submitted 2017-02-01; First posted 2017-03-03 (Actual); Results first posted 2021-12-03 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Human Immunodeficiency Virus; Depression
Keywords: HIV; Medication adherence; PMTCT; Depression
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Depression; Medication Adherence | interventions — Inhalation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: INSPireD (Experimental): This 5-8 session group intervention, "Integrating Nuanced Support for Perinatal adherence and Depression", aimed to decrease depressive symptoms and improve antiretroviral adherence among HIV-infected pregnant and postpartum women. Intervention content was based on two established cognitive-behavioral interventions: problem-solving therapy and Cognitive Behavioral Therapy for Adherence and Depression.
  Interventions: Behavioral: Integrating Nuanced Support for Perinatal adherence and Depression
- Treatment-as-usual + abbreviated intervention (Other): This group received treatment-as usual, plus the option of completing an abbreviated version of the intervention (one session of problem-solving related to adherence and mental health) at the conclusion of study.
  Interventions: Behavioral: Integrating Nuanced Support for Perinatal adherence and Depression

INTERVENTIONS:
Behavioral: Integrating Nuanced Support for Perinatal adherence and Depression — A 5-8 session intervention to decrease depressive symptoms and improve antiretroviral adherence among HIV-infected pregnant and postpartum women
  Other Names: INSPireD

SUMMARY:
The main aim was to conduct a pilot field test of a group-based depression and adherence counseling intervention with HIV-infected women in the perinatal period. Participants were HIV-infected women living in KwaZulu-Natal, South Africa.

DETAILED DESCRIPTION:
The main aim of this study was to conduct a pilot field test of a group-based counseling intervention with HIV-infected women in the perinatal period as delivered by a lay counselor. The primary goal of the intervention was to reduce symptoms of perinatal depression and increase adherence to antiretroviral therapy among HIV-infected women during pregnancy and the postpartum period.

ELIGIBILITY:
Inclusion Criteria:

* Currently pregnant
* HIV-infected and diagnosed with HIV during the index pregnancy
* Meet criteria for a major depressive episode
* Currently on antiretroviral therapy
* Receiving antenatal care at PMMH Gateway clinic
* Primary language English or isiZulu
* Access to a phone and willing to give researchers permission to reach them via phone
* Resident of Umlazi

Exclusion Criteria:

* Unable or unwilling to provide informed consent
* Active untreated, major mental illness (untreated psychosis, bipolar disorder, dementia, or active suicidality) that would interfere with study participation
* Less than 18 years of age

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2016-11-09 (Actual); Primary Completion 2017-03-24 (Actual); Study Completion 2017-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Psaros, PhD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- Massachusetts General Hospital, Boston, Massachusetts, United States
- MatCH Research, Durban, South Africa

REFERENCES:
- [Background] Lu M, Safren SA, Skolnik PR, Rogers WH, Coady W, Hardy H, Wilson IB. Optimal recall period and response task for self-reported HIV medication adherence. AIDS Behav. 2008 Jan;12(1):86-94. doi: 10.1007/s10461-007-9261-4. Epub 2007 Jun 19. PMID 17577653
- [Derived] Psaros C, Stanton AM, Raggio GA, Mosery N, Goodman GR, Briggs ES, Williams M, Bangsberg D, Smit J, Safren SA. Optimizing PMTCT Adherence by Treating Depression in Perinatal Women with HIV in South Africa: A Pilot Randomized Controlled Trial. Int J Behav Med. 2023 Feb;30(1):62-76. doi: 10.1007/s12529-022-10071-z. Epub 2022 Mar 8. PMID 35260947
- [Derived] Choi KW, Smit JA, Coleman JN, Mosery N, Bangsberg DR, Safren SA, Psaros C. Mapping a Syndemic of Psychosocial Risks During Pregnancy Using Network Analysis. Int J Behav Med. 2019 Apr;26(2):207-216. doi: 10.1007/s12529-019-09774-7. PMID 30805768

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between November 9, 2016 and March 3, 2017 from a district antenatal clinic in KwaZulu Natal, South Africa.
Groups:
- Intervention: INSPireD: This 5-8 session, group-based intervention, "Integrating Nuanced Support for Perinatal Adherence and Depression", had three primary goals: (1) improving adherence to ART during pregnancy and the postpartum period; (2) planning for contraceptive use; and (3) improving depressive symptoms among HIV-infected pregnant and postpartum women. Intervention content was based on two established cognitive-behavioral interventions: problem-solving therapy and CBT for adherence and depression.The intervention was delivered by a trained lay counselor, who completed a five-day training on counseling skills and intervention content, and received bi-monthly clinical supervision throughout the study.
- Treatment-as-usual + Abbreviated Intervention: The control group received treatment-as usual (standard of care counseling services), plus the option of completing an abbreviated version of the intervention (i.e., one session of problem-solving related to adherence and depression) at the conclusion of study.
Period: Overall Study
Arm/Group | Intervention: INSPireD | Treatment-as-usual + Abbreviated Intervention
Started | 14 | 9
Post-Treatment Assessment | 12 | 6
Completed | 8 | 2
Not Completed | 6 | 7
Not completed — Lost to Follow-up | 2 | 0
Not completed — Reason Unknown | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Intervention: INSPireD: This 5-8 session group intervention, "Integrating Nuanced Support for Perinatal adherence and Depression", aimed to decrease depressive symptoms and improve antiretroviral adherence among HIV-infected pregnant and postpartum women. Intervention content was based on two established cognitive-behavioral interventions: problem-solving therapy and CBT for adherence and depression.
- Control: Treatment-as-usual + Abbreviated Intervention: The control group received treatment-as usual, plus the option of completing an abbreviated version of the intervention (one session of problem-solving related to adherence and mental health) at the conclusion of study.
- Total: Total of all reporting groups
Arm/Group | Intervention: INSPireD | Control: Treatment-as-usual + Abbreviated Intervention | Total
Number analyzed (Participants) | 14 | 9 | 23
Age, Continuous [Median (Full Range); unit: years] | 25 [19 to 37] | 24 [18 to 32] | 24 [18 to 37]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 9 | 23
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 14 | 9 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 9 | 23
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Africa | 14 | 9 | 23
Highest Level of Schooling [Count of Participants; unit: Participants]
  Up to Grade 12 | 8 | 5 | 13
  Incomplete Post-Secondary | 5 | 4 | 9
  Complete Post-Secondary | 1 | 0 | 1
Current Employment Status [Count of Participants; unit: Participants]
  Not Employed | 10 | 6 | 16
  Full-Time Employed | 2 | 2 | 4
  Part-Time Employed | 2 | 1 | 3
Monthly Income [Count of Participants; unit: Participants]
  0-499 RAND | 3 | 2 | 5
  500-999 RAND | 0 | 1 | 1
  1000-1999 RAND | 1 | 2 | 3
  2000-2999 RAND | 0 | 1 | 1
  3000-3999 RAND | 0 | 2 | 2
  4000-4999 RAND | 2 | 1 | 3
  5000+ RAND | 4 | 0 | 4
  Don't know | 4 | 0 | 4
Trying to Get Pregnant [Count of Participants; unit: Participants]
  Yes, trying to get pregnant | 1 | 2 | 3
  No, not trying to get pregnant | 13 | 7 | 20
In a Relationship with Father of Current Pregnancy [Count of Participants; unit: Participants]
  No | 0 | 1 | 1
  Yes | 14 | 8 | 22
Partner's HIV Status [Count of Participants; unit: Participants]
  HIV Positive | 5 | 3 | 8
  HIV Negative | 0 | 1 | 1
  Don't know | 9 | 5 | 14

OUTCOME MEASURES:

1. Primary Outcome: Adherence to Antiretroviral Therapy Per Self-Report
Description: Adherence to ART during the previous month was measured through a composite score developed by Lu et al. (2008). The composite score combines the scores of three items into a single self-reported adherence score; the three items assess medication use frequency, percentage of time that the medication was taken as prescribed, and a rating of one's ability to take prescribed medication. The percent item had 11 response categories (0, 10, 20…100%), whereas the frequency and ability items had six response categories that were assigned scores of 0, 20, 40, 60, 80, and 100, with 100 considered to be perfect adherence.
Time Frame: Baseline, Post-Treatment (8-10 weeks), 3-Month Follow-Up (up to 6 months post-baseline)
Population: In the intervention arm, 14 participants completed a baseline assessment, 12 completed a post-treatment assessment, and 9 completed a three-month follow-up assessment. In the control arm, 9 participants completed a baseline assessment, 6 completed a post-treatment assessment, and 2 completed a three-month follow-up assessment.
Measure: Mean (Standard Deviation); unit: percentage of self-reported adherence
Arm/Group | Intervention: INSPireD | Control: Treatment-as-usual + Abbreviated Intervention
Number analyzed (Participants) | 14 | 9
percentage of self-reported adherence
  Baseline | 85.3 (12.9) | 79.0 (14.0)
  Post-Treatment: number analyzed (Participants) | 12 | 6
  Post-Treatment | 92.8 (8.7) | 77.8 (15.4)
  3-Month Follow-Up: number analyzed (Participants) | 8 | 2
  3-Month Follow-Up | 88.7 (9.3) | 89.2 (5.9)
Statistical Analysis 1: Comparison: Intervention: INSPireD vs Control: Treatment-as-usual + Abbreviated Intervention; Test type: Superiority — Conducted at post-treatment time point; p = 0.11, Mixed Models Analysis
Statistical Analysis 2: Comparison: Intervention: INSPireD vs Control: Treatment-as-usual + Abbreviated Intervention; Test type: Superiority — Conducted at 3-month follow-up time point; p = 0.56, Mixed Models Analysis

2. Primary Outcome: Adherence to Antiretroviral Therapy Per MEMS Caps
Description: Objective ART adherence data were collected using the Medication Event Monitoring System (MEMS), which comprises a pill bottle with a digitized cap that measures and records when the bottle was opened each day. MEMS timepoints were defined as average MEMS use across the two-week period prior to each of the three assessment visits.
Time Frame: Baseline, Post-Treatment (8-10 weeks), 3-Month Follow-Up (up to 6 months post-baseline)
Population: Sixteen participants (12 intervention, 4 control) were included in the MEMS analysis at baseline, 12 (10 intervention, 2 control) were included at post-treatment, and 7 (6 intervention, 1 control) were included at 3-month follow-up. Data for 7 participants were not included at baseline due to: inconsistent use or non-use (n=2), lost to follow-up (n=4), and relocated (n=1).Three were excluded from final analyses due to broken caps or consistent cap non-use over the three measurement periods.
Measure: Mean (Standard Deviation); unit: percentage of MEMS-recorded adherence
Arm/Group | Intervention: INSPireD | Control: Treatment-as-usual + Abbreviated Intervention
Number analyzed (Participants) | 12 | 4
percentage of MEMS-recorded adherence
  Baseline | 99.4 (2.2) | 92.9 (14.3)
  Post-Treatment: number analyzed (Participants) | 10 | 2
  Post-Treatment | 98.6 (3.0) | 100.0 (0.0)
  3-Month Follow-Up: number analyzed (Participants) | 6 | 1
  3-Month Follow-Up | 92.8 (6.4) | 85.7 (NA) — MEMS data were available for only 1 participant from the control arm at the 3-month follow-up timepoint.
Statistical Analysis 1: Comparison: Intervention: INSPireD vs Control: Treatment-as-usual + Abbreviated Intervention; Test type: Superiority — Main effect for time calculated at 3-month follow-up time point; p < 0.05, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; Fixed effects coefficient (β) = -12.7, 95% CI 2-sided [-22.29 to -3.15]

3. Primary Outcome: Level of Depressive Symptoms Per Edinburgh Postnatal Depression Scale (EPDS)
Description: The 10-item Edinburgh Postnatal Depression Scale (EPDS) was used to measure depressive symptoms at baseline, post-treatment, and three-month follow-up; higher scores indicate more severe depressive symptoms. The minimum possible score is 0, and maximum score is 30. A standard clinical cutoff of 13 on the EPDS was used to distinguish women with and without probable depression.
Time Frame: Baseline, Post-Treatment (8-10 weeks), 3-Month Follow-Up (up to 6 months post-baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention: INSPireD | Control: Treatment-as-usual + Abbreviated Intervention
Number analyzed (Participants) | 14 | 9
score on a scale
  Baseline | 20.8 (5.7) | 20.3 (6.1)
  Post-Treatment: number analyzed (Participants) | 12 | 6
  Post-Treatment | 1.2 (1.7) | 11.8 (9.0)
  3-Month Follow-Up: number analyzed (Participants) | 8 | 2
  3-Month Follow-Up | 2.1 (2.9) | 6.5 (9.2)
Statistical Analysis 1: Comparison: Intervention: INSPireD vs Control: Treatment-as-usual + Abbreviated Intervention; Test type: Superiority — Interaction evaluated at post-treatment time point; p < 0.005, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; Fixed effects coefficient (β) = -11.1, 95% CI 2-sided [-18.41 to -3.83]
Statistical Analysis 2: Comparison: Intervention: INSPireD vs Control: Treatment-as-usual + Abbreviated Intervention; Test type: Superiority — Main effect for time at 3-month follow-up time point; p < 0.005, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; Fixed effects coefficient (β) = -13.8, 95% CI 2-sided [-22.50 to -5.17]

4. Primary Outcome: Number of Participants With Depressive Symptoms Per MINI - Meeting Criteria for MDD
Description: Current and past major depressive disorder was measured using the 17-item Major Depressive Episode Module of the Mini International Neuropsychiatric Interview (MINI). If an individual indicates either that they were "consistently depressed or down, most of the day, nearly every day for the past two weeks" or that they were "less interested in doing most things or less able to enjoy the things that they used to enjoy most of the time," they are asked about 7 symptoms of depression. To meet criteria for a current major depressive episode, at least three symptoms must be endorsed.
Time Frame: Baseline, Post-Treatment (8-10 weeks), 3-Month Follow-Up (up to 6 months post-baseline)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention: INSPireD | Control: Treatment-as-usual + Abbreviated Intervention
Number analyzed (Participants) | 14 | 9
Participants
  Baseline | 12 | 7
  Post-Treatment: number analyzed (Participants) | 12 | 6
  Post-Treatment | 0 | 2
  3-Month Follow-Up: number analyzed (Participants) | 8 | 2
  3-Month Follow-Up | 0 | 1

5. Secondary Outcome: Level of Stigma Per HIV/AIDS Stigma Instrument (HASI-P)
Description: HIV-related stigma was measured at baseline, post-treatment, and 3-month follow-up using the HIV/AIDS Stigma Instrument - People Living with AIDS (HASI-P). Three sub-scales from the full scale were used: negative self-perception (5 items), social isolation (5 items), and verbal abuse (8 items). Responses are rated on a four-point Likert scale from "never" (0) to "most of the time" (3). Subscale score ranges were 0-15 (negative self-perception and social isolation) and 0-24 (verbal abuse); subscale scores were summed to compute a total score (range 0-54). Higher scores indicate higher levels of stigma.
Time Frame: Baseline, Post-Treatment (8-10 weeks), 3-Month Follow-Up (up to 6 months post-baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention: INSPireD | Control: Treatment-as-usual + Abbreviated Intervention
Number analyzed (Participants) | 14 | 9
score on a scale
  Baseline | 14.3 (10.2) | 24.3 (12.6)
  Post-Treatment: number analyzed (Participants) | 12 | 6
  Post-Treatment | 6.3 (10.2) | 12.8 (10.9)
  3-Month Follow-Up: number analyzed (Participants) | 8 | 2
  3-Month Follow-Up | 2.5 (6.7) | 12.5 (17.7)
Statistical Analysis 1: Comparison: Intervention: INSPireD vs Control: Treatment-as-usual + Abbreviated Intervention; Test type: Superiority — Main effect for condition; p < 0.05, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; Fixed effects coefficient (β) = -10.1, 95% CI 2-sided [-19.58 to -0.67]
Statistical Analysis 2: Comparison: Intervention: INSPireD vs Control: Treatment-as-usual + Abbreviated Intervention; Test type: Superiority — Main effect for time at post-treatment time point; p < 0.01, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; Fixed effects coefficient (β) = -12.8, 95% CI 2-sided [-22.14 to -3.37]

6. Secondary Outcome: Level of Social Support Per Duke-UNC Functional Social Support Questionnaire
Description: Social support was assessed using a modified version of the Duke-UNC Functional Social Support Questionnaire, a 10-item scale evaluating availability of emotional, informational, and tangible support. Items are rated on a 4-point Likert scale; number of persons providing support is also assessed. The maximum possible score is 40 and minimum score is 0; higher scores indicate greater perceived social support.
Time Frame: Baseline, Post-Treatment (8-10 weeks), 3-Month Follow-Up (up to 6 months post-baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention: INSPireD | Control: Treatment-as-usual + Abbreviated Intervention
Number analyzed (Participants) | 14 | 9
score on a scale
  Baseline | 33.9 (5.8) | 27.7 (9.6)
  Post-Treatment: number analyzed (Participants) | 12 | 6
  Post-Treatment | 35.3 (5.6) | 28.0 (4.5)
  3-Month Follow-Up: number analyzed (Participants) | 8 | 2
  3-Month Follow-Up | 36.4 (5.5) | 36.5 (3.5)
Statistical Analysis 1: Comparison: Intervention: INSPireD vs Control: Treatment-as-usual + Abbreviated Intervention; Test type: Superiority — Main effect for condition; p < 0.05, Mixed Models Analysis — The threshold for statistical significance was p = 0.05; Fixed effects coefficient (β) = 6.2, 95% CI 2-sided [0.50 to 11.88]

ADVERSE EVENTS:
Time Frame: Up to 6 months post-baseline
Arm/Group | Intervention: INSPireD | Control: Treatment-as-usual + Abbreviated Intervention
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/9
Other Adverse Events (participants affected / at risk) | 0/14 | 0/9

LIMITATIONS AND CAVEATS:
(1) The small sample size in this study limited our ability to detect consistent statistically significant differences between arms. (2) High baseline adherence likely impacted our ability to detect differences between study arms. (3) Session scheduling was an additional and substantial challenge. While women were largely able to complete most planned sessions, this required flexibility on the part of the interventionist, and all but precluded a group meeting format.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-25): https://cdn.clinicaltrials.gov/large-docs/17/NCT03069417/Prot_SAP_000.pdf